CLINICAL TRIAL: NCT00434811
Title: Islet Transplantation in Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CIT-07
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Insulin dependence; Hypoglycemia; Hypoglycemia unawareness
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Antilymphocyte Serum; Sirolimus; Tacrolimus; Etanercept; Islets of Langerhans Transplantation; Basiliximab; prolactin-binding protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Islet Transplantation (Experimental): Participants will receive up to three separate islet transplants and a regimen of immunosuppressive medications consisting of antithymocyte globulin (ATG), sirolimus, and low-dose tacrolimus.
  Interventions: Biological: Allogeneic Pancreatic Islet Cells; Biological: Antithymocyte Globulin; Drug: Sirolimus; Drug: Tacrolimus; Biological: Etanercept; Procedure: Islet Transplantation; Biological: Basiliximab

INTERVENTIONS:
Biological: Allogeneic Pancreatic Islet Cells — 200 ml suspension of allogenic human purified islets
Biological: Antithymocyte Globulin — Participants will begin receiving ATG 2 days prior to the first islet transplant. ATG will continue to be given until Day 2 post-transplant.
Drug: Sirolimus — Participants will begin receiving sirolimus 2 days prior to the first islet transplant and will be given for the duration of the study.
  Other Names: Rapamycin
Drug: Tacrolimus — On Day 1 post-transplant, participants will receive tacrolimus, which will also be taken for the duration of the study.
  Other Names: FK-506; Fujimycin
Biological: Etanercept — Etanercept will be taken on the day of transplant and Days 3, 7, and 10 post-transplant.
Procedure: Islet Transplantation — Transplantation of pancreatic islet cell
Biological: Basiliximab — Basiliximab will be used in place of ATG for the second and third transplants, if they are necessary.
  Other Names: chimeric mouse-human antiCD25; Ig gamma-1 chain C region

SUMMARY:
Type 1 diabetes is an autoimmune disease in which the insulin-producing pancreatic beta cells are destroyed, resulting in poor blood sugar control. The purpose of this study is to determine the safety and effectiveness of islet transplantation, combined with immunosuppressive medications, for treating type 1 diabetes in individuals experiencing hypoglycemia unawareness and severe hypoglycemic episodes.

DETAILED DESCRIPTION:
Type 1 diabetes is commonly treated with the administration of insulin, either by multiple insulin injections or by a continuous supply of insulin through a wearable pump. Insulin therapy allows long-term survival in individuals with type 1 diabetes; however, it does not guarantee constant normal blood sugar control. Because of this, long-term type 1 diabetic survivors often develop vascular complications, such as diabetic retinopathy, an eye disease that can cause poor vision and blindness, and diabetic nephropathy, a kidney disease that can lead to kidney failure. Some individuals with type 1 diabetes develop hypoglycemia unawareness, a life-threatening condition that is not easily treatable with medication and is characterized by reduced or absent warning signals for hypoglycemia. For such individuals, transplantation of pancreatic islets is a possible treatment option. Unfortunately, insulin independence among islet transplant recipients tends to decline over time. New strategies aimed at promoting engraftment of transplanted islets are needed to improve the clinical outcomes associated with this procedure. The purpose of this study is determine the safety and efficacy of islet transplantation, when combined with an immunosuppressive medication regimen, for treating type 1 diabetes in individuals experiencing hypoglycemia unawareness and severe hypoglycemic episodes. This study will also seek to improve the understanding of determinants of success and failure of islet transplants for type 1 diabetes.

Eligible participants will be randomly assigned to this study or a site-specific Phase 2 islet transplantation study. Participants in this study will receive up to three separate islet transplants and a regimen of immunosuppressive medications consisting of antithymocyte globulin (ATG), sirolimus, and low-dose tacrolimus.

Transplantations will involve an inpatient hospital stay and infusion of islets into a branch of the portal vein. Participants who do not achieve or maintain insulin independence by Day 75 post-transplant will be considered for a second islet transplant. Participants who remain dependent on insulin for longer than 1 month after the second transplant and who show partial graft function will be considered for a third islet transplant. Basiliximab will be used in place of ATG for the second and third transplants, if they are necessary. Participants who do not meet the criteria for a subsequent transplant and do not have a functioning graft will enter a reduced follow-up period.

There will be up to 19 study visits following each transplant. A physical exam, review of adverse events, and blood collection will occur at most visits. A chest x-ray, abdominal ultrasound, electrocardiogram, quality of life questionnaires, urine collection, and glomerular filtrating rate (GFR) testing will occur at some visits. Participants will also test their own blood glucose levels at least five times per day throughout the study. A 24-month follow-up period will take place after the participant's last transplant.

ELIGIBILITY:
Inclusion Criteria:

* Mentally stable and able to comply with study procedures
* Clinical history compatible with type 1 diabetes with onset of disease at less than 40 years of age, insulin dependence for at least 5 years at study entry, and a sum of age and insulin dependent diabetes duration of at least 28
* Absent stimulated C-peptide (less than 0.3 ng/ml) 60 and 90 minutes post-mixed-meal tolerance test
* Involvement of intensive diabetes management, defined as:

  1. Self-monitoring of glucose values no less than a mean of three times each day averaged over each week
  2. Administration of three or more insulin injections each day or insulin pump therapy
  3. Under the direction of an endocrinologist, diabetologist, or diabetes specialist with at least three clinical evaluations during the past 12 months prior to study enrollment
* At least one episode of severe hypoglycemia in the past 12 months, defined as an event with one of the following symptoms: memory loss; confusion; uncontrollable behavior; irrational behavior; unusual difficulty in awakening; suspected seizure; seizure; loss of consciousness; or visual symptoms, compatible with hypoglycemia in which the individual required assistance of another subject was unable to treat him/herself person and which was associated with either a blood glucose level less than 54 mg/dl or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration in the 12 months prior to study enrollment
* Reduced awareness of hypoglycemia. More information about this criterion, including specific definition of hypoglycemia unawareness, is in the protocol.

Exclusion Criteria:

* Body mass index (BMI) greater than 30 kg/m2 or weight less than or equal to 50 kg
* Insulin requirement of more than 1.0 IU/kg/day or less than 15 U/day
* HbA1c greater than 10%
* Untreated proliferative diabetic retinopathy
* Systolic blood pressure higher than 160 mmHg or diastolic blood pressure higher than 100 mmHg
* Measured glomerular filtration rate using iohexol of less than 80 ml/min/1.73mm2. More information about this criterion is in the protocol.
* Presence or history of macroalbuminuria (greater than 300 mg/g creatinine)
* Presence or history of panel-reactive anti-HLA antibody levels greater than background by flow cytometry. More information about this criterion is in the protocol.
* Pregnant, breastfeeding, or unwilling to use effective contraception throughout the study and 4 months after study completion
* Presence or history of active infection, including hepatitis B, hepatitis C, HIV, or tuberculosis.
* Negative for Epstein-Barr virus by IgG determination
* Invasive aspergillus, histoplasmosis, or coccidioidomycosis infection in the past year
* History of malignancy except for completely resected squamous or basal cell carcinoma of the skin
* Known active alcohol or substance abuse
* Baseline Hgb below the lower limits of normal, lymphopenia, neutropenia, or thrombocytopenia
* History of Factor V deficiency
* Any coagulopathy or medical condition requiring long-term anticoagulant therapy after transplantation or individuals with an INR greater than 1.5
* Severe coexisting cardiac disease, characterized by any one of the following conditions:

  1. Heart attack within the last 6 months
  2. Evidence of ischemia on functional heart exam within the year prior to study entry
  3. Left ventricular ejection fraction less than 30%
* Persistent elevation of liver function tests at the time of study entry
* Symptomatic cholecystolithiasis
* Acute or chronic pancreatitis
* Symptomatic peptic ulcer disease
* Severe unremitting diarrhea, vomiting, or other gastrointestinal disorders that could interfere with the ability to absorb oral medications
* Hyperlipidemia despite medical therapy, defined as fasting LDL cholesterol greater than 130 mg/dl (treated or untreated) and/or fasting triglycerides greater than 200 mg/dl
* Currently receiving treatment for a medical condition that requires chronic use of systemic steroids except for the use of 5 mg or less of prednisone daily, or an equivalent dose of hydrocortisone, for physiological replacement only
* Treatment with any antidiabetic medication other than insulin within the past 4 weeks
* Use of any study medications within the past 4 weeks
* Received a live attenuated vaccine(s) within the past 2 months
* Any medical condition that, in the opinion of the investigator, might interfere with safe participation in the trial

  * Treatment with any immunosuppressive regimen at the time of enrollment.
  * A previous islet transplant.
  * A previous pancreas transplant, unless the graft failed within the first week due to thrombosis, followed by pancreatectomy and the transplant occurred more than 6 months prior to enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-10; Primary Completion 2012-09 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with a HbA1c less than 7.0% AND free of severe hypoglycemic events | From Day 28 to Day 365 (inclusive) following the first islet transplant, with the day of transplant designated Day 0
  The proportion of participants with HbA1c ≤7.0% AND free of severe hypoglycemic events from Day 28 to Day 365 inclusive, following the first islet transplant, with the day of transplant designated Day 0.

SECONDARY OUTCOMES:
Percent reduction in insulin requirements | 75 days following the first and subsequent islet transplant
HbA1c on Day 75 Status Post the First and Subsequent Islet Transplant | 75 days following the first and subsequent islet transplant
  The target level for HbA1c for this study is 7.0%. This value is the level recommended by the American Diabetes Association and is considered to be the clinically relevant goal for subjects with Type 1 diabetes (T1D). A HbA1c level of 6.5% is the goal recommended by the American College of Endocrinology.
Mean amplitude of glycemic excursions (MAGE) | 75 days following the first and subsequent islet transplant
  A MAGE >11.1 mmol/L (200 mg/dL) is indicative of marked glycemic lability.
Glycemic liability index (LI) | 75 days following the first and subsequent islet transplant
Ryan hypoglycemia severity score (HYPO) | 75 days following the first and subsequent islet transplant
Basal (fasting) and 90-minute glucose and C-peptide derived from mixed meal tolerance test (MMTT) | 75 days following the first and subsequent islet transplant
β-score on Day 75 Status Post the First and Subsequent Islet Transplant | 75 days following the first and subsequent islet transplant
  Beta-score: an assessment of beta-cell function after islet transplantation.
C-peptide:glucose creatinine ratio | 75 days following the first and subsequent islet transplant
Acute insulin response to glucose, insulin sensitivity, and disposition index derived from the insulin-modified frequently sampled intravenous glucose tolerance (FSIGT) test | 75 days following the first and subsequent islet transplant
Glucose variability and hypoglycemia duration derived from the continuous glucose monitoring system (CGMS) | 75 days following the first and subsequent islet transplant
Assessment of Quality of Life Using the Short Form 36 Health Survey: Day 75 Status Post First and Final Islet Transplant | 75 days following the first and subsequent islet transplant
  The Short-Form 36 Health Survey (SF-36®) is comprised of 36 items and 2 component scores, the Physical Component Score and the Mental Component Score. Each component is transformed into a 0-100 scale (higher numbers indicate greater quality of life) and normalized to have a mean of 50 and standard deviation of 10 for the 1998 general US population. SF-36 results unit of measure: Units on a Scale.
Incidence of worsening retinopathy | 365 days following the first islet transplant
Proportion of insulin-independent Participants on Day 365 Status Post the First and Final Islet Transplant | 365 days following the first and final islet transplant
Percent reduction in insulin requirements | 365 days following the first and final islet transplant
HbA1c on Day 365 Status Post the First and Final Islet Transplant | 365 days following the first and final islet transplant
  The target level for HbA1c for this study is 7.0%. This value is the level recommended by the American Diabetes Association and is considered to be the clinically relevant goal for subjects with Type 1 diabetes (T1D). A HbA1c level of 6.5% is the goal recommended by the American College of Endocrinology.
MAGE | 365 days following the first and final islet transplant
  A MAGE >11.1 mmol/L (200 mg/dL) is indicative of marked glycemic lability.
Glycemic liability index (LI): Day 365 Status Post First and Final Islet Transplant | 365 days following the first and final islet transplant
Clarke score | 365 days following the first and final islet transplant
  The Clarke survey provides a composite indices of hypoglycemia frequency, severity, and symptom recognition.
HYPO score | 365 days following the first and final islet transplant
  The HYPO(glycemia) score provides a composite indices of hypoglycemia frequency, severity, and symptom recognition.
Basal (fasting) and 90-minute glucose and C-peptide (MTT) | 365 days following the first and final islet transplant
β-score on Day 365 Status Post First and Final Islet Transplant | 365 days following the first and final islet transplant
  Beta-score: an assessment of beta-cell function after islet transplantation.
C-peptide: glucose creatinine ratio | 365 days following the first and final islet transplant
Assessment of Quality of Life Using the Short Form 36 Health Survey: Day 365 Status Post First and Final Islet Transplant | 365 days following the first and final islet transplant
  The Short-Form 36 Health Survey (SF-36®) is comprised of 36 items and 2 component scores, the Physical Component Score and the Mental Component Score. Each component is transformed into a 0-100 scale (higher numbers indicate greater quality of life) and normalized to have a mean of 50 and standard deviation of 10 for the 1998 general US population. SF-36 results unit of measure: Units on a Scale.
Proportion of participants receiving a second islet transplant | 365 days following the first and final islet transplant
Proportion of participants receiving a third islet transplant | 365 days following the first and final islet transplant
Incidence and severity of adverse events related to the islet transplant procedure | 75 days following each transplant and 365 days following the first and final islet transplant
Incidence and severity of adverse events related to the immunosuppression therapy | 75 days following each transplant and 365 days following the first and final islet transplant
Incidence of a change in the immunosuppression drug regimen | 75 days following each transplant and 365 days following the first and final islet transplant
Incidence of immune sensitization defined by detecting anti-HLA antibodies not present prior to transplantation | 75 days following each transplant and 365 days following the first and final islet transplant
Proportion of insulin-independent participants on Day 75 Status Post First and Subsequent Islet Transplant | 75 days following first and subsequent islet transplant
Acute insulin response to glucose insulin sensitivity, and disposition index derived from the FSIGT test | 365 days following the first and final islet transplant
  Frequently Sampled Intravenous Glucose Tolerance (FSIGT), a measure of insulin-independence, a clinically relevant measure of islet graft function.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Hering, MD, Study Chair — University of Minnesota; Olle Korsgren, PhD, Study Chair — Uppsala University Hospital; Ali Naji, PhD, Study Chair — University of Pennsylvania; Camillo Ricordi, MD, Study Chair — University of Miami; James Shapiro, MD, PhD, Study Chair — University of Alberta; Andrew Posselt, MD, PhD, Study Chair — University of California, San Francisco; Nicole Turgeon, MD, Study Chair — Emory University; Xunrong Luo, MD, PhD, Study Chair — Northwestern Univerity
Locations (8):
- United States (7):
  - University of Callifornia, San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Participant level data access and additional relevant materials are available to researchers and the public at: https://www.immport.org/home.
  The study Identifier in ImmPort is SDY1178.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data is available. ImmPort is a long-term archive of clinical and mechanistic data.
Access Criteria: Register for ImmPort at: https://www.immport.org/registration and submit a rationale for the purpose of requesting study data access.
  ImmPort is a long-term archive of clinical and mechanistic data, a National Institute of Allergy and Infectious Diseases Division of Allergy, Immunology and Transplantation (NIAID DAIT)-funded data repository. This archive is in support of the NIH mission to share data with the public. Data shared through ImmPort is provided by NIH-funded programs, other research organizations and individual scientists, ensuring these discoveries will be the foundation of future research.
URL: https://www.immport.org/home

REFERENCES:
- [Background] Shapiro AM, Ricordi C, Hering BJ, Auchincloss H, Lindblad R, Robertson RP, Secchi A, Brendel MD, Berney T, Brennan DC, Cagliero E, Alejandro R, Ryan EA, DiMercurio B, Morel P, Polonsky KS, Reems JA, Bretzel RG, Bertuzzi F, Froud T, Kandaswamy R, Sutherland DE, Eisenbarth G, Segal M, Preiksaitis J, Korbutt GS, Barton FB, Viviano L, Seyfert-Margolis V, Bluestone J, Lakey JR. International trial of the Edmonton protocol for islet transplantation. N Engl J Med. 2006 Sep 28;355(13):1318-30. doi: 10.1056/NEJMoa061267. PMID 17005949
- [Background] Harlan DM. Islet Transplantation for Hypoglycemia Unawareness/Severe Hypoglycemia: Caveat Emptor. Diabetes Care. 2016 Jul;39(7):1072-4. doi: 10.2337/dci16-0008. No abstract available. PMID 27330121
- [Result] Rickels MR, Liu C, Shlansky-Goldberg RD, Soleimanpour SA, Vivek K, Kamoun M, Min Z, Markmann E, Palangian M, Dalton-Bakes C, Fuller C, Chiou AJ, Barker CF, Luning Prak ET, Naji A. Improvement in beta-cell secretory capacity after human islet transplantation according to the CIT07 protocol. Diabetes. 2013 Aug;62(8):2890-7. doi: 10.2337/db12-1802. Epub 2013 Apr 29. PMID 23630300
- [Result] Hering BJ, Clarke WR, Bridges ND, Eggerman TL, Alejandro R, Bellin MD, Chaloner K, Czarniecki CW, Goldstein JS, Hunsicker LG, Kaufman DB, Korsgren O, Larsen CP, Luo X, Markmann JF, Naji A, Oberholzer J, Posselt AM, Rickels MR, Ricordi C, Robien MA, Senior PA, Shapiro AM, Stock PG, Turgeon NA; Clinical Islet Transplantation Consortium. Phase 3 Trial of Transplantation of Human Islets in Type 1 Diabetes Complicated by Severe Hypoglycemia. Diabetes Care. 2016 Jul;39(7):1230-40. doi: 10.2337/dc15-1988. Epub 2016 Apr 18. PMID 27208344
- [Result] Ricordi C, Goldstein JS, Balamurugan AN, Szot GL, Kin T, Liu C, Czarniecki CW, Barbaro B, Bridges ND, Cano J, Clarke WR, Eggerman TL, Hunsicker LG, Kaufman DB, Khan A, Lafontant DE, Linetsky E, Luo X, Markmann JF, Naji A, Korsgren O, Oberholzer J, Turgeon NA, Brandhorst D, Chen X, Friberg AS, Lei J, Wang LJ, Wilhelm JJ, Willits J, Zhang X, Hering BJ, Posselt AM, Stock PG, Shapiro AM, Chen X. National Institutes of Health-Sponsored Clinical Islet Transplantation Consortium Phase 3 Trial: Manufacture of a Complex Cellular Product at Eight Processing Facilities. Diabetes. 2016 Nov;65(11):3418-3428. doi: 10.2337/db16-0234. Epub 2016 Jul 27. PMID 27465220
- [Derived] Foster ED, Bridges ND, Feurer ID, Eggerman TL, Hunsicker LG, Alejandro R; Clinical Islet Transplantation Consortium. Improved Health-Related Quality of Life in a Phase 3 Islet Transplantation Trial in Type 1 Diabetes Complicated by Severe Hypoglycemia. Diabetes Care. 2018 May;41(5):1001-1008. doi: 10.2337/dc17-1779. Epub 2018 Mar 21. PMID 29563196
- [Derived] Senior PA, Bellin MD, Alejandro R, Yankey JW, Clarke WR, Qidwai JC, Schwieger TR, Eggerman TL, Robien MA, Rickels MR; Clinical Islet Transplantation Consortium. Consistency of quantitative scores of hypoglycemia severity and glycemic lability and comparison with continuous glucose monitoring system measures in long-standing type 1 diabetes. Diabetes Technol Ther. 2015 Apr;17(4):235-42. doi: 10.1089/dia.2014.0289. Epub 2015 Jan 28. PMID 25629445
- [Derived] Gala-Lopez B, Kin T, O'Gorman D, Pepper AR, Senior P, Humar A, Shapiro AM. Microbial contamination of clinical islet transplant preparations is associated with very low risk of infection. Diabetes Technol Ther. 2013 Apr;15(4):323-7. doi: 10.1089/dia.2012.0297. Epub 2013 Feb 25. PMID 23438305
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- Available data/document: Study Protocol: SDY1178 — http://www.immport.org/immport-open/public/home/studySearch — ImmPort study ID is SDY1178.
- Available data/document: Complete set of descriptive data and results: SDY1178 — http://www.immport.org/immport-open/public/home/studySearch — ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts. This archive is in support of the NIH mission to share data with the public.